CLINICAL TRIAL: NCT01842776
Title: Care Transitions in Renal Disease Patients
Acronym: CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fresenius Medical Care North America (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20129159
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this pilot is to reduce the 30-day hospital readmission rate for dialysis patients. It is a quality improvement project that consistent of 4 "tracks." Tracks 1 & 2: Implement use of checklists of activities for staff to complete when patients are admitted to the hospital, and post-hospitalization with emphasis on fluid assessment, nutrition management, patient coaching, and communication between institutions. Track 3: Work with physicians to develop process to individualize post-hospitalization dialysis orders and improve medication reconciliation. Track 4: Use a renal Care Transitions Case Manager to follow patients in the hospital and 30 days post-hospitalization to facilitate care and patient coaching.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients
* All patients admitted to the hospital during the study period

Exclusion Criteria:

* Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hemodialysis patients
Sampling Method: Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
30-day readmission rate | Participants will be followed for the duration of each hospital stay and 30 days post-hospitalization, for an expected average of 37 days.
  Number of hospitalizations that occur within 30 days after discharge from an initial index hospitalization (convert to percentage of 30-day readmissions).

CONTACTS AND LOCATIONS:
Locations (1):
- Fresenius, Franklin, Tennessee, United States